CLINICAL TRIAL: NCT03915769
Title: A Phase 2/3, Multicenter, Randomized, Double-blind, Placebo-controlled Study of Oral Ozanimod to Evaluate Efficacy and Long-term Safety in Japanese Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: To Evaluate Efficacy and Long-term Safety of Ozanimod in Japanese Subjects With Moderately to Severely Active Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RPC01-3103; U1111-1230-3228 (Registry Identifier: WHO)
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Colitis, Ulcerative
Keywords: Ulcerative colitis; Ozanimod; colitis; Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative; Colitis; Ulcer | interventions — ozanimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- 0.46 mg ozanimod oral capsule once daily (QD) (Experimental): It will be a 7-day dose escalation regimen in the IP consisting of 4 days of treatment with 0.23 mg ozanimod, followed by 3 days of treatment with 0.46 mg ozanimod, followed by 0.46 mg ozanimod.
  Interventions: Drug: Ozanimod
- 0.92 mg ozanimod oral capsule QD (Experimental): It will be a 7-day dose escalation regimen in the IP consisting of 4 days of treatment with 0.23 mg ozanimod, followed by 3 days of treatment with 0.46 mg ozanimod, followed by 0.92 mg ozanimod.
  Interventions: Drug: Ozanimod
- Placebo oral capsule QD (Placebo Comparator): It will be a 7-day dose escalation regimen in the IP consisting of 4 days of treatment with a placebo capsule, followed by 3 days of treatment with two placebo capsules, followed by two placebo capsules.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ozanimod — Ozanimod is an orally bioavailable, small molecule compound that activates the sphingosine 1-phosphate 1 receptor (S1P1) and the S1P 5 receptor (S1P5), although it is more selective towards S1P1 over S1P5
  Arms: 0.46 mg ozanimod oral capsule once daily (QD); 0.92 mg ozanimod oral capsule QD
Other: Placebo — The placebo is a capsule that contains no study medication but looks exactly like the study medication capsule.
  Arms: Placebo oral capsule QD

SUMMARY:
Japanese patients with moderate or severe active ulcerative colitis as a subject when ozanimod 0.46 mg or 0.92 mg is orally administered is evaluated about dose response, efficacy and safety with placebo as a control.

DETAILED DESCRIPTION:
Following the up to 5-week Screening Period, eligible subjects will be randomized to enter the 12 weeks placebo-controlled Induction Period (IP). Subjects who are responders at Week 12 will continue on their assigned treatment in the 40-week Maintenance Period (MP). Non responders at Week 12 have the option to enter the Open-label Extension (OLE). Subjects who complete the MP will be given the option to participate in the OLE. Subjects that enter the MP and experience disease relapse will also have the option to enter the OLE. The OLE will continue until marketing launch (about 4 years of ozanimod for Ulcerative colitis (UC), or until the Sponsor discontinues the development program.

ELIGIBILITY:
Inclusion Criteria:

Main Inclusion Criteria for Induction and Maintenance Periods

1. Subject is a Japanese male or female subjects aged 18 to 75 years at the time of signing the informed consent form (ICF) at Screening.
2. Subject has had Ulcerative Colitis (UC) diagnosed at least 3 months prior to first investigational product administration. The diagnosis should be confirmed by clinical and endoscopic evidence and corroborated by a histopathology report.
3. Subject has evidence of UC extending ≥ 15 cm from the anal verge as determined by Baseline endoscopy (flexible sigmoidoscopy or colonoscopy).
4. Subject has active UC defined as Mayo score of 6 to 12 inclusive, with endoscopic subscore of ≥ 2, a rectal bleeding score of ≥ 1, and a stool frequency score ≥ 1.

Main Inclusion Criteria for Open-label Extension Period

Subjects must satisfy the following criteria to be enrolled in the study:

1. Must have completed the Week 12 Visit and is non-responder at Week 12
2. Who completes the IP and enters the MP, completes participation through the last study treatment visit at Week 52 with maintaining clinical response, OR experiences disease relapse during the MP

Exclusion Criteria:

Main Exclusion Criteria

1. Subject has severe extensive colitis
2. Subject has diagnosis of Crohn's disease or indeterminate colitis or the presence or history of a fistula consistent with Crohn's disease or microscopic colitis or radiation colitis or ischemic colitis.
3. Subject has positive stool examination for pathogens (ova and parasites, bacteria) or positive test for toxin producing Clostridium difficile (C. difficile) at Screening.4. Subject is pregnant or breastfeeding

5. Subject has clinically relevant cardiovascular conditions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with clinical response | At Week 12
  Defined as a reduction from Baseline in the complete Mayo score of ≥ 3 points and ≥ 30%, and a reduction from Baseline in the rectal bleeding subscore of ≥ 1 point or an absolute rectal bleeding subscore of ≤ 1 point

SECONDARY OUTCOMES:
Proportion of subjects with clinical remission | At Week 12 and Week 52
  Defined as: Definition 1. Complete Mayo score of ≤ 2 points with no individual subscore of > 1 point, Definition 2. Rectal bleeding subscore = 0 and stool frequency subscore ≤ 1 (and a decrease of ≥ 1 point from the Baseline stool frequency subscore) and endoscopy subscore ≤ 1
Proportion of subjects with a clinical response | At Week 12 and Week 52
  Defined as a reduction from Baseline in the 9-point Mayo score of ≥ 2 points and ≥ 35%, and a reduction from Baseline in the rectal bleeding subscore of ≥ 1 point or an absolute rectal bleeding subscore of ≤ 1 point
Proportion of subjects with endoscopic improvement | At Week 12 and Week 52
  Defined as an endoscopy subscore of ≤ 1 point
Proportion of subjects with mucosal healing | At Week 12 and Week 52
  Defined as an endoscopy subscore of ≤ 1 point and a Geboes index score < 2.0
Proportion of subjects with a clinical response | At Week 9
  Defined as a reduction from Baseline in the partial Mayo score of ≥ 2 points and ≥ 30%, and a reduction from Baseline in the rectal bleeding subscore of ≥ 1 point or an absolute rectal bleeding subscore of ≤ 1 point
Change in the EuroQol-5 Dimension (EQ-5D) from baseline | At Week 12
  Is a quality of life questionnaires and will be collected from all subjects at visits
Proportion of subject with clinical response | At week 52
  Defined as a reduction from Baseline in the complete Mayo score of ≥ 3 points and ≥ 30%, and a reduction from Baseline in the rectal bleeding subscore of ≥ 1 point or an absolute rectal bleeding subscore of ≤ 1 point
Proportion of subjects in remission while off corticosteroids for any length of time | Up to week 52
  Proportion of subjects in remission while off corticosteroids for any length of time
Adverse Event (AE) | From enrollment until at least 75 days after completion of study treatment
  Number of participants with adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (67):
- Japan (67):
  - Local Institution - 104, Sapporo, Hokkaido
  - Local Institution - 105, Nishinomiya, Hyōgo
  - Local Institution - 156, Okayama, Okayama-ken
  - Local Institution - 153, Osaka, Osaka
  - Local Institution - 132, Osaka, Osaka-shi
  - Local Institution - 131, Iruma-gun, Saitama
  - Local Institution - 138, Bunkyo-ku, Tokyo
  - Local Institution - 139, Abiko
  - Local Institution - 152, Aki-gun
  - Local Institution - 122, Chikushino-shi
  - Local Institution - 150, Fujiidera
  - Local Institution - 114, Fukui
  - Local Institution - 124, Fukui
  - Local Institution - 161, Fukuoka
  - Local Institution - 164, Fukuoka
  - Local Institution - 155, Fukuoka
  - Local Institution - 140, Gifu
  - Local Institution - 151, Hakodate
  - Local Institution - 133, Hirosaki
  - Local Institution - 160, Hiroshima
  - Local Institution - 106, Hiroshima
  - Local Institution - 126, Hitachi, Ibaraki
  - Local Institution - 162, Iizuka
  - Local Institution - 134, Isehara City, Kanagawa
  - Local Institution - 120, Kahoku-gun
  - Local Institution - 135, Kannonji
  - Local Institution - 101, Kashihara
  - Local Institution - 158, Kashiwa
  - Local Institution - 157, Kawagoe
  - Local Institution - 163, Kobe
  - Local Institution - 130, Kobe
  - Local Institution - 121, Komatsu
  - Local Institution - 144, Kōriyama
  - Local Institution - 142, Kurume
  - Local Institution - 165, Kurume
  - Local Institution - 111, Kurume, Fukuoka
  - Local Institution - 141, Kyoto
  - Local Institution - 118, Matsuyama
  - Local Institution - 108, Minatoku
  - Local Institution - 107, Minatoku
  - Local Institution - 109, Mitaka
  - Local Institution - 110, Morioka
  - Local Institution - 125, Nagaoka
  - Local Institution - 167, Nagoya
  - Local Institution - 136, Okayama
  - Local Institution - 127, Osaki-shi
  - Local Institution - 119, Ōgaki
  - Local Institution - 159, Ōita
  - Local Institution - 113, Ōtsu
  - Local Institution - 154, Saga
  - Local Institution - 116, Saitama
  - Local Institution - 145, Sakai
  - Local Institution - 102, Sakura
  - Local Institution - 103, Sapporo
  - Local Institution - 147, Sapporo
  - Local Institution - 146, Sendai
  - Local Institution - 128, Shinagawa-ku, Tokyo
  - Local Institution - 117, Shinjuku
  - Local Institution - 137, Shizuoka
  - Local Institution - 149, Sunto-gun
  - Local Institution - 112, Takamatsu
  - Local Institution - 115, Takatsuki
  - Local Institution - 143, Takatsuki
  - Local Institution - 166, Toshima-ku
  - Local Institution - 129, Toyama
  - Local Institution - 123, Tsu
  - Local Institution - 148, Utsunomiya

IPD SHARING:
Plan to Share IPD: Yes
https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com